CLINICAL TRIAL: NCT03533244
Title: A Multicenter, Prospective, Randomized, Double-Masked, Phase 2 Study Evaluating the Safety, Tolerability, and Efficacy of Topical AG-86893 in Patients With Pterygium
Brief Title: A Study of the Response to AG-86893 in Patients With Pterygium Hyperemia
Acronym: SURPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allgenesis Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2-86893-001
Record Dates: First submitted 2018-04-27; First posted 2018-05-23 (Actual); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-01

CONDITIONS: Pterygium
Keywords: Hyperemia
MeSH Terms: conditions — Pterygium; Hyperemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle Eye Drops (Placebo Comparator): One drop, three times daily to the study eye for 28 days
  Interventions: Drug: Vehicle Eye Drops
- 0.1% AG-86893 Eye Drops (Experimental): One drop, three times daily to the study eye for 28 days
  Interventions: Drug: 0.1% AG-86893 Eye Drops
- 0.3% AG-86893 Eye Drops (Experimental): One drop, three times daily to the study eye for 28 days
  Interventions: Drug: 0.3% AG-86893 Eye Drops

INTERVENTIONS:
Drug: 0.1% AG-86893 Eye Drops — One drop, three times daily to the study eye for 28 days
  Arms: 0.1% AG-86893 Eye Drops
Drug: 0.3% AG-86893 Eye Drops — One drop, three times daily to the study eye for 28 days
  Arms: 0.3% AG-86893 Eye Drops
Drug: Vehicle Eye Drops — One drop, three times daily to the study eye for 28 days
  Arms: Vehicle Eye Drops

SUMMARY:
A pterygium is a wing-shaped, benign tissue growth which forms on the surface of the conjunctiva and grows towards the cornea. It can eventually lead to vision impairment. The precise cause of pterygium formation is unknown but new blood vessel growth and fibroblastic structures are characteristics of the disease. AG-86893 is an eye drop being developed to treat hyperemia (redness) and growth of the pterygium.

Hypothesis

1. AG-86893 dosed three times daily for 28 consecutive days has an acceptable safety profile as measured by the incidence and severity of adverse events (AEs) compared with vehicle
2. At least 1 concentration of AG-86893 is effective, as measured by the mean change from baseline in conjunctival hyperemia (redness), compared with vehicle

ELIGIBILITY:
Inclusion Criteria:

* Good health with no clinically significant findings based on the medical history, electrocardiogram, vital signs, blood chemistry, hematology, and urinalysis findings, as determined by the investigator
* Females of childbearing potential must have a negative pregnancy test at baseline and must be on established, adequate contraception and males must use condoms if their partner is of childbearing potential and their female partner should also use an additional effective means of contraception, or they must agree to abstain from sexual intercourse with a female partner for the duration of the study; contraception should be continued for 3 months after the last dose.
* Presence of pterygium with associated conjunctival hyperemia (redness) of grade ≥2 as assessed by a central reading center.

Exclusion Criteria:

* History or presence of any ocular diseases other than pterygium or its sequelae (after-effects), including neoplasia (uncontrolled overgrowth)
* Diagnosis of ocular hypertension or glaucoma requiring use of intraocular pressure-lowering medication
* Use of contact lenses during the study in the study eye
* History or evidence of ocular surgeries in the study eye at any time
* History of liver dysfunction or current abnormal liver enzymes
* Pregnancy, plans for pregnancy, or breastfeeding during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - M.T. Coroneo Pty Ltd, Randwick, New South Wales
  - H2Vision Centre, Sippy Downs, Queensland
  - Bendigo Eye Clinic, Bendigo, Victoria
  - Essendon Eye Clinic, Essendon, Victoria
  - The Geelong Eye Centre, Waurn Ponds, Victoria
  - Lions Eye Institute, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle Eye Drops | 0.1% AG-86893 Eye Drops | 0.3% AG-86893 Eye Drops
Started | 20 | 22 | 22
Completed | 18 | 21 | 22
Not Completed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Eye Drops | 0.1% AG-86893 Eye Drops | 0.3% AG-86893 Eye Drops | Total
Number analyzed (Participants) | 20 | 22 | 22 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.4) | 54.7 (11.9) | 49.0 (10.7) | 51.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 11 | 26
  Male | 10 | 17 | 11 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 18 | 21 | 19 | 58
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 20 | 22 | 22 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Conjunctival Hyperemia Score
Description: Assessed by digital ocular photography; each quadrant of the eye (superior, inferior, nasal, temporal) will be scored using a 5-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe) and graded by a reading center. The overall conjunctival score is the average of the four quadrants. Assessments are made by subtracting the score at Baseline from the score on Day 28. An increase in value indicates worsening of hyperemia, while a decrease indicates improvement.
Time Frame: Baseline and Day 28
Population: modified intent-to-treat (mITT)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle Eye Drops | 0.1% AG-86893 Eye Drops | 0.3% AG-86893 Eye Drops
Number analyzed (Participants) | 18 | 22 | 22
score on a scale | -0.056 (0.120) | -0.330 (0.109) | -0.352 (0.109)
Statistical Analysis 1: Comparison: Vehicle Eye Drops vs 0.3% AG-86893 Eye Drops; An empirical sample size estimation was used as this was an exploratory study. The null hypothesis is that there is no difference between AG-86893 and AG-86893 Vehicle. It is expected that the active group is at least 50% better than the vehicle; Test type: Superiority; p = 0.218, Mixed Models Analysis — To reserve the family-wise error rate, the main treatment effect will be first assessed at the global level at alpha = 0.05. If this is significant, then pairwise comparisons will be conducted using the Bonferroni adjustment for multiplicity
Statistical Analysis 2: Comparison: Vehicle Eye Drops vs 0.1% AG-86893 Eye Drops; Test type: Superiority; p = 0.290, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in Conjunctival Hyperemia Score in the Quadrant With the Pterygium
Description: Assessed by digital ocular photography; the quadrant with the pterygium will be scored using a 5-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe) and graded by a reading center. Assessments are made by subtracting the score at Baseline from the score on Day 28. An increase in value indicates worsening of hyperemia, while a decrease indicates improvement.
Time Frame: Baseline and Day 28
Population: Per protocol (PP)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle Eye Drops | 0.1% AG-86893 Eye Drops | 0.3% AG-86893 Eye Drops
Number analyzed (Participants) | 18 | 21 | 22
score on a scale | -0.111 (0.153) | -0.429 (0.142) | -0.500 (0.138)
Statistical Analysis 1: Comparison: Vehicle Eye Drops vs 0.3% AG-86893 Eye Drops; Test type: Superiority; p = 0.193, Mixed Models Analysis
Statistical Analysis 2: Comparison: Vehicle Eye Drops vs 0.1% AG-86893 Eye Drops; Test type: Superiority; p = 0.399, Mixed Models Analysis

3. Post Hoc Outcome: Percent of Patients With a 1-point Decrease in Hyperemia Score in the Quadrant With the Pterygium
Description: Assessed by digital ocular photography; the quadrant with the pterygium will be scored using a 5-point scale and graded by a reading center. A 1-point reduction in hyperemia score is considered clinically meaningful.
Time Frame: Day 28
Population: Per protocol (PP)
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Eye Drops | 0.1% AG-86893 Eye Drops | 0.3% AG-86893 Eye Drops
Number analyzed (Participants) | 18 | 21 | 22
Participants | 3 | 11 | 12
Statistical Analysis 1: Comparison: Vehicle Eye Drops vs 0.3% AG-86893 Eye Drops; Test type: Superiority; p = 0.015, Fisher Exact
Statistical Analysis 2: Comparison: Vehicle Eye Drops vs 0.1% AG-86893 Eye Drops; Test type: Superiority; p = 0.022, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each patient until Day 84 (exit).
Arm/Group | Vehicle Eye Drops | 0.1% AG-86893 Eye Drops | 0.3% AG-86893 Eye Drops
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 5/20 | 5/22 | 15/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Eye Drops (N=20) | 0.1% AG-86893 Eye Drops (N=22) | 0.3% AG-86893 Eye Drops (N=22)
Conjunctival Discoloration (Eye disorders) | 0 | 1 | 10
Vision blurred (Eye disorders) | 1 | 1 | 4
Dry eye (Eye disorders) | 0 | 0 | 2
Eye pruritis (Eye disorders) | 1 | 2 | 0
Eye pain (Eye disorders) | 1 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Episcleritis (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 2 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Influenza (Ear and labyrinth disorders) | 1 | 0 | 0
Nasopharyngitis (Ear and labyrinth disorders) | 1 | 0 | 0
Pneumonia (Ear and labyrinth disorders) | 1 | 0 | 0
Viral upper respiratory tract infection (Ear and labyrinth disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT03533244/SAP_000.pdf
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT03533244/Prot_002.pdf